CLINICAL TRIAL: NCT05559216
Title: The Effect of Upper Extremity Plyometric Exercises on Proprioception, Time to Peak Torque and Performance in Young Female Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Çağla MELEP, Physiotherapist, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1185180
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Plyometric Exercise; Proprioception; Upper Quarter y Balance Test; The Closed Kinetic Chain Upper Extremity Stability Test
Keywords: plyometric exercise; upper extremity; proprioception; upper quarter y balance test; basketball; ckcuest
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basketball Players (Other)
  Interventions: Other: Plyometric Training

INTERVENTIONS:
Other: Plyometric Training — Plyometric training exercises are being given to the participants to see the changes after the 8 week period

SUMMARY:
Plyometric exercises are used in many sports branches to increase sportive performance and neuromuscular coordination. It is known that side values such as the time to reach peak torque next to muscle strength, which is one of the evaluations of sportive performance, are also important. Our aim with this study is; To evaluate the effects of plyometric exercises on proprioception, time to peak torque and performance in young female basketball players by training the dominant and non-dominant upper extremity on these parameters.

DETAILED DESCRIPTION:
Basketball is one of the most popular indoor games in the world, played in almost every region without exception. It includes skillful movement that includes shooting, defense and dribbling. Compared to other team sports, the main differences demanded by basketball players during training and matches are faster and shorter accelerations and decelerations, explosive deflections, jumps, and various potentially traumatic contacts between players. a basketball shot; consists of preparation, raising the ball, stability, release and follow-up. During overhead sports, the shoulder must accept the high joint loads produced by the lower extremity and trunk and efficiently transfer this energy to the upper extremity along the kinetic chain. The articulations of the shoulder complex provide a range of motion for the shoulder joint and allow complex movements such as throwing. This mobility depends on the controlled and synchronized movement of the shoulder joints. Shoulder flexion prior to ball release has been reported to be an important factor for increasing ball release height. Plyometric exercises are drills or exercises that aim to combine shear strength with explosive reactive movement type. Plyometric exercises involve rapid stretching (i.e. lengthening) of a muscle just before a rapid concentric contraction. This combined action is commonly referred to as the stretch-shorten cycle (SSC). Pre-stretching is the most important stage of plyometric activity, because it increases the excitability of neurological receptors, which increases the reactivity of the neuromuscular system. Swanik et al. suggested that plyometric activities may facilitate neural adaptations that increase proprioception, kinesthesia, and muscle performance characteristics. The ability to rapidly generate torque is an important skill in most athletic studies, and it has been suggested that assessment of muscle recruitment patterns in athletes (such as time to peak torque) provides better indicators of functional performance than assessment of peak torque alone. Sudden movements in the joints require a rapid muscle contraction capacity to stabilize it. Parameters such as acceleration time and time to peak torque have been established in the literature as muscle recruitment variables that provide valuable information regarding neuromuscular readiness to produce maximal contractions. The time to peak torque (in milliseconds), reflecting muscle coordination, is defined as the time from initial contraction to peak torque during muscle contraction. Therefore, TPT data can be used synonymously with contraction time. In a previous study using upper extremity plyometric exercises, an 8-week training consisting of 3 days a week warm-up and cool-down periods was deemed appropriate. Considering the above information, our aim with this study is; To evaluate the effects of plyometric exercises on proprioception, time to peak torque and performance in young female basketball players by training the dominant or non-dominant upper extremity on these parameters.

Evaluations of our thesis work will be carried out in the Laboratories of Istanbul Medical Faculty, Department of Sports Medicine. The research will be carried out only in the Laboratories of the Istanbul Faculty of Medicine, Department of Sports Medicine and no other Center will be used. The number of research centers is 1. Although it is planned to start the research on 01.09.2022 in the event that an Ethics Committee is taken, it is planned to be completed by 09.01.2023.

Working method ; Young female basketball players will be divided into 2 equal groups as dominant arm exercise group and non-dominant arm exercise group after the tests done in the clinic. Then they will do the given exercises as instructed. The same evaluations will be repeated when they come back to the clinic at the end of 8 weeks.

Evaluations to be applied in the study:

* Obtaining demographic information: Age, height, weight, dominant leg, previous injuries, how long he has been involved in this sport,
* Pre- and post-exercise proprioception and strength measurements using Cybex Humac NORM
* For functional performance evaluation; Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) and Upper Quarter Y Balance Test (UQYBT) are planned to be applied in a laboratory environment.
* Note the time to reach peak torque during the force test for later comparison

The work plan:

It is planned to start our thesis study in March after the approval of the ethics committee. It is planned that the evaluations will be completed within 2 weeks, the exercise training to be applied will last for 6 weeks, then the same evaluations will be made and the same will continue for 2 weeks. It is foreseen that the first evaluation dates will be between 09.01.2022-01.06.2023, exercise training will be between 09.01.2022-11.01.2022, and the second evaluation date will be between 11.01.2022-12.01.2023. Our study is planned to last for 6 months.

Experimental stages: For exercise training to individuals; -Seven plyometric upper extremity exercises (2 sets, 15 repetitions) will be planned for the athletes 3 times a week for 8 weeks.

Exercises :

* Arm swings (fexion, extension and across the body)
* D1 D2 pnf patterns (with elastic band)
* Punching (with 1kg dumbbells)
* IR and ER with elastic band
* Overhead throws
* Reverse catches
* Push-up (knees on the ground) Shoulder stretches will be performed for warm-up and cool-down periods before and after the exercise program.

Proprioception measurement with Cybex Isokinetic Dynanometer will be done for the evaluation of the athlete before and after the exercise program.

-UQYBT and CKCUEST tests will be used for evaluation before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* signing the Informed Voluntary Consent form by agreeing to participate in the study voluntarily
* Being a young female basketball player
* Have not had a shoulder injury in the past six months

Exclusion Criteria:

* Having an existing upper extremity injury
* Having an upper extremity injury in the last 6 months
* Complaints of pain in manual strength test

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Proprioception | 8 weeks
  The player will be laying down on the Cybex Humac NORM device and the investigators will be quetioning the player to put her arm in the same position as the investigatorsdo while her eyes are closed. The investigators will show the player 3 times and make he player do the angles themselves again 3 times and note down the degrees that are more than ours or less ( eg. if the investigators show them 90° and they do 93° the investigators write down the 3°.) The angles the investigators are using are 0°, 90° and 172°. After the exercise period ends, same staff will measure the same angles and see if there is any difference.
Time To Peak Torque | 8 weeks
  Before and after changes in participants time to peak torque times

SECONDARY OUTCOMES:
Performance | 8 weeks
  The performance tests the investigators are using are the Upper Quarter Y Balance Test and The Closed Kinetic Chain Upper-Extremity Stability Test (CKCUEST). With upper quarter Y balance test the investigators are aiming to measure players' balance, proprioception, strength, and greater range of motion. The Closed Kinetic Chain Upper-Extremity Stability Test (CKCUEST) is an objective, easy functional test that can be used to measure components of muscle performance of the shoulder complex in a closed-kinetic chain position and places high demands on its stabilizers. The investigators again test our players on these before and after the 8 weeks period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No